CLINICAL TRIAL: NCT06008184
Title: Real-time Monitoring of Cortisol - Comparison of Cortisol Levels in Four Biological Fluids
Acronym: SensoCort
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Principal Investigator, Nelly Pitteloud, Professor, Centre Hospitalier Universitaire Vaudois
Other Study IDs: CER-VD : 2021-01674
Record Dates: First submitted 2023-08-18; First posted 2023-08-23 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Adrenal Insufficiency; Cushing Syndrome; Hyperaldosteronism
MeSH Terms: conditions — Adrenal Insufficiency; Cushing Syndrome; Hyperaldosteronism | interventions — Blood Specimen Collection; Sweating

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy controls
  Interventions: Other: 24 hours sampling of 4 biological fluids (blood, ISF, sweat and saliva); Other: 24 hours sampling of ISF or sweat (after validating the correlation with blood)

INTERVENTIONS:
Other: 24 hours sampling of 4 biological fluids (blood, ISF, sweat and saliva) — 24 hours sampling of 4 biological fluids:
  * blood: sampling every 20 minutes (through a venous catheter)
  * ISF: automated sampling every 20 minutes (microdialysis technique connected to U-Rhythm device)
  * Sweat : collection of 1 to 3 samples at 4 differents timepoints
  * Saliva : sampling every hour (except during the night)
Other: 24 hours sampling of ISF or sweat (after validating the correlation with blood) — 24 hours sampling in an ambulatory setting

SUMMARY:
Cortisol is an essential for life hormone secreted in a pulsatile pattern on a diurnal rhythm. Given the complexity of cortisol secretion on a circadian rhythm with pulsations, current methods of cortisol measurement have limitations.

Therefore, a non-invasive and ambulatory method would be useful to measure cortisol levels in real-time.

The main aim of the study is to compare cortisol levels across biological fluids (sweat, saliva, interstitial fluid, and blood) in order to validate in the long term a continuous and non-invasive cortisol measurement device (currently under development).

ELIGIBILITY:
Healthy controls:

Inclusion Criteria:

* age between 18 and 30 years old
* normal BMI 18 to 25 kg/m2
* weight stability

Exclusion Criteria:

* pregnancy, breastfeeding, irregular menses
* any medical treatment
* any medical issues
* pilocarpine allergy, or latex allergy
* glaucoma or acute irritis

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy volunteers
Sampling Method: Probability Sample
Enrollment: 12 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Cortisol levels in 4 biologicals fluids | 24 hours
  Comparison of cortisol levels in these 4 biological fluids

SECONDARY OUTCOMES:
Aldosterone levels in 4 biological fluids | 24 hours
  Comparison of aldosterone levels in these 4 biological fluids
Glucocorticoid - comparison of repeated measures of glucocorticoid concentrations (cortisol, 18OHF, cortisone) profiles - over a period of 24 hours | 24 hours
  Study of the diurnal rhythm and pulsatility in healthy participants (and later patients)
  * Diurnal rhythm: cosinor analysis. Comparison of nadir/acme of cortisol concentrations (and 18OHF, cortisone) among participants. Amplitude of the curve
  * Pulsatility analysis: frequency of the pulses and amplitude
Mineralocorticoid - comparison of repeated measures of aldosterone concentrations profiles - over a period of 24 hours | 24 hours
  Study of the diurnal rhythm and pulsatility in healthy participants (and later patients)
  * Diurnal rhythm: cosinor analysis. Comparison of nadir/acme of aldosterone concentrations among participants. Amplitude of the curve
  * Pulsatility analysis: frequency of the pulses and amplitude

CONTACTS AND LOCATIONS:
Overall Officials: Nelly Pitteloud, MD, Principal Investigator — Centre Hospitalier Universitaire Vaudois
Locations (1):
- Centre Hospitalier Universitaire Vaudois (CHUV), Lausanne, Canton of Vaud, Switzerland